CLINICAL TRIAL: NCT00251368
Title: Multicenter Study of 9-AC in Refractory Leukemia
Brief Title: Multicenter Study of 9-Aminocamptothecin (9-AC) in Patients With Refractory Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94-115
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Leukemia, Myelocytic, Acute; Acute Lymphocytic Leukemia
Keywords: leukemia; 9-Aminocamptothecin; AML; ALL; refractory leukemia; relapsed leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — 9-aminocamptothecin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 9-Aminocamptothecin (9-AC)

SUMMARY:
The purpose of this study is to evaluate the side effects of 9-Aminocamptothecin (9-AC) and to determine the best dose which should be used to treat leukemia.

DETAILED DESCRIPTION:
* The treatment patients will receive involves a continuous infusion of 9-AC intravenously for a 72 hour period. Since we are unsure of the safest and most effective dose, successive groups of 4-7 patients will receive larger doses of this drug until the largest dose given safely is established.
* Prior to the start of therapy a bone marrow aspirate and biopsy will be taken for diagnostic and research purposes. A bone marrow exam will be repeated at 48 hours in order to determine the effects of 9-AC on leukemic cells in the bone marrow. A bone marrow scan will also be performed 14 days after the start of therapy to assess response.
* Frequent blood testing will be done throughout treatment, including blood samples to determine the levels of the 9-AC in the blood.
* Treatment could be stopped prematurely if any of the following occur: 1) drug causes severe side effects, 2) the drug does not control the leukemia, or 3) the doctors or the patient feel that it is no longer in the patients best interest to receive this therapy.
* Approximately 7 days after the conclusion of the 9-AC infusion, it is likely that the patient's blood counts will be low and will require support with antibiotics, red cell transfusions and platelet transfusions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* AML or ALL in first or subsequent relapse, secondary AML, or CML in blastic phase
* Central venous access
* ECOG performance status of less than or equal to 2
* Bilirubin < 1.3
* SGOT < 2 x ULN
* Alkaline phosphatase < 2 x ULN
* Creatinine < 1.5

Exclusion Criteria:

* Undergone bone marrow transplantation
* Uncontrolled infection
* Other active malignancy
* HIV positivity
* Serious medical or psychiatric illness
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 1995-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the toxicity and maximum tolerated dose of 9-AC administered as a 72 hour infusion in patients with relapsed/refractory leukemia. | Years

SECONDARY OUTCOMES:
To analyze the pharmacokinetics in these patients. | years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stone, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts